CLINICAL TRIAL: NCT00303576
Title: A Phase I/II Double-Blind, Randomized Study of the Safety, Tolerability and Systemic Absorption of TMC120 Vaginal Microbicide Gel and Matching Placebo in Healthy HIV-Negative Women.
Brief Title: A Safety and Tolerability Study of Dapivirine (TMC120) Vaginal Microbicide Gel
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: International Partnership for Microbicides, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IPM003
Record Dates: First submitted 2006-03-15; First posted 2006-03-17 (Estimated); Last update posted 2006-07-31 (Estimated); Status verified 2006-07

CONDITIONS: HIV Infections
Keywords: HIV-1; HIV Seronegativity
MeSH Terms: conditions — HIV Infections | interventions — Dapivirine; Vaginal Creams, Foams, and Jellies

INTERVENTIONS:
Drug: dapivirine (TMC120) vaginal gel

SUMMARY:
Approximately 112 HIV-negative women, aged 18 to 50, will be enrolled in this multicenter study at four sites. Volunteers will be randomized to dapivirine (TMC120) vaginal gel or matching placebo gel. The volunteers will receive investigational product for a total of 42 days. Volunteers will be monitored on days 7, 28 and 42 for safety, tolerability and compliance.

ELIGIBILITY:
Inclusion Criteria:

* HIV-negative
* Willing to participate and sign an informed consent
* Willing to be tested for HIV, use an experimental vaginal gel, and to be randomized to a study group that includes the possibility of being assigned to a placebo group.
* Willing to use two forms of contraception during the study.
* Willing to undergo pelvic examinations with colposcopy and photographic documentation according to the protocol throughout the study.
* Have a regular menstrual cycle defined as having a minimum of 21 days and a maximum of 36 days between menses.
* Willing to abstain from using any vaginal product (other than the study product or placebo).
* Willing to be sexually abstinent from randomization until completion of Day 7 evaluations.

Exclusion Criteria:

* Currently pregnant or breast-feeding.
* Clinically detectable genital abnormality on the vulva, vaginal walls or cervix.
* Laboratory confirmed gonorrhea, chlamydia, trichomonas, syphilis, or vaginal candidiasis or clinically diagnosed genital ulcer disease or active HSV-2 lesions.
* Breakthrough bleeding or gynecologic surgery within 60 days prior to randomization.
* Symptomatic bacterial vaginosis and unwilling to undergo treatment.
* Women who require treatment for tuberculosis (TB) within 21 days prior to randomization.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 112
Dates: Start 2005-10; Study Completion 2006-07

PRIMARY OUTCOMES:
Local and systemic safety and tolerability.

CONTACTS AND LOCATIONS:
Overall Officials: Zeda Rosenberg, ScD, Study Director — Beijing Immupeutics Medicine Technology Limited
Locations (4):
- Projet Ubuzima, Kigali, Rwanda
- South Africa (2):
  - Reproductive Health Research Unit - Sheshisani IPM Clinic, Yeoville, Johannesburg
  - Farmovs-Parexel, Bloemfontein
- Kilimanjaro Reproductive Health Program, Moshi, Tanzania